CLINICAL TRIAL: NCT00613093
Title: Phase II Trial of Temodar Plus O6-Benzylguanine (O6-BG) (NSC 637037) in the Treatment of Patients With Temodar-Resistant Malignant Glioma
Brief Title: Ph. II Temozolomide + O6-BG in Treatment of Pts w Temozolomide-Resistant Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Keryx / AOI Pharmaceuticals, Inc. (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4260
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2012-11

CONDITIONS: Glioblastoma Multiforme; Anaplastic Glioma
Keywords: Temodar; Temozolomide; O6-BG; O6-Benzylguanine; NSC 637037; Temodar-Resistant Malignant Glioma; Brain tumor; CNS tumor; Cerebral glioblastoma; Anaplastic astrocytomas; Glioma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Central Nervous System Neoplasms; Astrocytoma; Glioma | interventions — Temozolomide; O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with glioblastoma multiforme (Active Comparator)
  Interventions: Drug: Temodar and O6-Benzylguanine (BG)
- Patients with Anaplastic Glioma (Active Comparator)
  Interventions: Drug: Temodar and O6-Benzylguanine (BG)

INTERVENTIONS:
Drug: Temodar and O6-Benzylguanine (BG) — Objectives of study are to define role of BG in restoring Temodar sensitivity in patients with Temodar-resistant malignant glioma and to further define the toxicity of combination therapy using Temodar + BG. 2 separate strata accrued independently of each other: Stratum 1-patients with glioblastoma multiforme (GBM). Stratum 2-patients with anaplastic glioma (AG).
  BG at 120mg/m2 administered intravenously over 1 hour followed immediately by 48-hour infusion at 30mg/m2/24 hours. Temodar 472mg/m2 administered orally, in fasting state, within 60 minutes of end of the 1-hour administration of BG infusion. Treatment cycles may be repeated every 28 days following dose of Temodar from previous cycle.
  Other Names: Temodar - Temozolomide; O6-Benzylguanine - O6-BG

SUMMARY:
Objectives:

To define role of O6-Benzylguanine (BG) in restoring Temodar (temozolomide) sensitivity in patients with Temodar-resistant malignant glioma.

To further define toxicity of combo therapy using Temodar + BG.

DETAILED DESCRIPTION:
2 separate strata accrued independently of each other: Stratum 1-patients with Glioblastoma Multiforme (GBM). Stratum 2-patients with Anaplastic Glioma [anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed (AA and AO)] .

BG at 120mg/m2 administered intravenously over 1 hour followed immediately by 48-hour infusion at 30mg/m2/24hrs. Temozolomide 472mg/m2 administered orally, in fasting state, within 60 minutes of end of the 1-hour administration of BG infusion. Treatment cycles may be repeated every 28 days following dose of Temodar from previous cycle.

Temodar has been well tolerated by both adults and children with most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea and vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, hepatotoxicity, anorexia, fatigue and hyperglycemia. Hypersensitivity reactions have not yet been noted with Temodar. As in the case with many anti-cancer drugs, Temodar may be carcinogenic. BG toxicities include agitation, lethargy, nausea, vomiting, rapid heart rate, elevated liver functions, & leukemia; but, not with BG as single agent. Transient lymphopenia has been seen with BG as single agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients have recurrent/progressive Malignant Glioma (MG). Stereotactic biopsy at time of recurrence/progression is only required if radiation-induced necrosis is suspected
* Patients have MG resistant to Temodar, which is defined as > or = to 25 percent increase in tumor growth on contrast enhanced MRI/CT within 8 weeks of last dose of Temodar
* Age > or = to 18 years
* Evidence of measurable enhancing disease on contrast-enhanced MRI, unless medically contraindicated.
* Interval of at least 2 weeks between prior surgical resection/ 4 weeks between prior radiotherapy/chemotherapy, and enrollment on protocol unless there is unequivocal evidence of tumor progression. However, patients treated with chemotherapy agents such as VP-16 who would normally be retreated after shorter intervals may be treated at usual starting time even if less than 4 weeks from last prior dose of chemotherapy
* Karnofsky performance score > or = to 60 percent
* Hematocrit > 29 percent, absolute neutrophil count (ANC) > 1,500 cells/microliter, platelets > 100,000 cells/microliter
* Serum creatinine <1.5 mg/dl, Blood Urea Nitrogen (BUN) <25 mg/dl, Serum Glutamic Oxaloacetic Transaminase (SGOT) & bilirubin <1.5 x upper limit of normal (ULN)
* For patients on corticosteroids, they must have been on stable dose for 1 week prior to entry, if clinically possible, and dose should not be escalated over entry dose level
* Signed informed consent approved by Institutional Review Board (IRB) prior to patient entry
* If sexually active, patients will take contraceptive measures for duration of treatments

Exclusion criteria:

* Pregnancy
* Co-medication that may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2002-10; Primary Completion 2006-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Radiographic evidence of tumor response | 6 months

SECONDARY OUTCOMES:
6 month progression-free survival | 6 months
Relationship between tumor AGT at original diagnosis & response to Temozolomide + O6-BG | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/